CLINICAL TRIAL: NCT01231022
Title: Study the Role of Stem Cell in Curing Drug Induced Liver Injury in Metastatic Breast Cancer
Brief Title: Study the Role of Stem Cell in Curing Drug Induced Liver Injury in Metastatic Breast Cancer (MBC)
Acronym: MBC
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Ren, Director, Peking University Cancer Hospital & Institute
Other Study IDs: DILI
Record Dates: First submitted 2010-10-20; First posted 2010-11-01 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
Keywords: breast neoplasm; Neoplasm Metastasis; Stem Cells; Drug-Induced Liver Injury
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — patients' blood sample
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators want to know the role of Peripheral hematopoietic stem cell infusion in avoiding Drug Induced Liver Injury,and also try to research SNPs genotyping associated with Drug Induced Liver Injury.

DETAILED DESCRIPTION:
1. The researcher investigate the incidence and the cause of Drug Induced Liver Injury in MBC.
2. Patients having a complete clinical history and physical examination, receive routine chemotherapy.
3. Venous blood Sample(4 ml)is collected before and after each cycle according to the planning time.
4. Genomic DNA,RNA and upper serum is isolated. ELISA、rt-PCR or PCR-direct sequencing is used to detect the protein or gene expression associated with liver function.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be histologically confirmed with metastatic breast cancer;
* an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Normal cardiac, hepatic, renal and bone marrow functions;
* Life expectancy ≥3 months;

Exclusion Criteria:

* previous history of other malignancies;
* Central nervous system metastases;
* Serious or uncontrolled concurrent medical illness.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: female patients with metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Protective effection of peripheral hematopoietic stem cell infusion for DILI | 3 months
  Patients receiving PHSC infusion after chemotherapy will have lower incidence of DILI. PHSC infusion may improve the liver function.

SECONDARY OUTCOMES:
SNPs genotyping associated with Drug Induced Liver Injury | 3 months
  Some SNPs will be find to associated with DILI.
Change of cytokines | 3 months
  Changes of cytokines in periphral blood related with liver function with be observed.

CONTACTS AND LOCATIONS:
Overall Officials: XU LIANG, MD and PhD, Principal Investigator — Peking University Cancer Hospital & Institute; JUN REN, MD and PhD, Study Chair — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China